CLINICAL TRIAL: NCT05833321
Title: Prospective Monocentric Study of the Detection of Sarcopenia in Clinical Practice in Patients With Ovarian or Endometrial Cancer Requiring Systemic Oncological Treatment
Brief Title: Prospective Study of Detection of Sarcopenia in Clinical Practice for Patient With Ovarian or Endometrial Cancer
Acronym: SARCO-GYN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHMS22005
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Neoplasms; Sarcopenia
MeSH Terms: conditions — Ovarian Neoplasms; Sarcopenia

STUDY DESIGN:
Intervention Model Description: prospective non-randomized interventional study
Masking Description: Inclusion criteria:
  * Patients at least 18 years old
  * Patient presenting with a diagnosis of cancer of ovarian origin with an indication for chemotherapy
  * Patient with a diagnosis of endometrial cancer with an indication for chemotherapy
  * Patient with no diagnosis of other types of cancer in the previous five years
  * Collection of consent
  * Patient affiliated to a Social Security scheme Non-inclusion criteria
  * Patient with cancer of ovarian origin not requiring chemotherapy treatment
  * Patient with endometrial cancer not requiring chemotherapy treatment
  * Discovery of an intercurrent cancer other than skin or cervix cancers.
  * Patient wearing a Pace maker
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventionnal (Experimental): "Hand Grip" Dynamometer Walk test SEFI Nutritional Intake Assessment Questionnaire
  Interventions: Diagnostic Test: Sarcopenia diagnostic test

INTERVENTIONS:
Diagnostic Test: Sarcopenia diagnostic test — measurement of impedance and physical tests ("hand grip" dynamometer, walking test), SEFI nutritional intake questionnaire

SUMMARY:
Prospective monocentric study, non-randomized of the detection of sarcopenia in clinical practice in patients with ovarian or endometrial cancer requiring systemic oncological treatment.

main question : Identify the criteria correlated with the presence of sarcopenia (defined by the measurement of the IMS by the CT-X method in L3) among the impedancemetry and the HAS malnutrition criteria.

Data collection will be done at 6 months, 12 months after the date of inclusion.

DETAILED DESCRIPTION:
Primary objective:Identify the criteria correlated to the presence of sarcopenia (defined by the measurement of the IMS by the CT-X method in L3) among the impedancemetry and the HAS malnutrition criteria

Main judgment criteria : Comparison between the groups of patients with sarcopenia (Morphometric measurement of the musculoskeletal surface index <39cm²/m² in L3 cross section) and without sarcopenia of the different evaluation criteria:

* Impedancemetry values:: muscle mass index in kg/m2 (IMS), fat-free mass in kg/m2 and metabolic activity index (phase angle)
* Percentage of weight loss
* BMI < 18.5 kg/m2
* Quantified reduction in muscle mass and/or function for patients < 70 years old
* Quantified reduction in muscle mass and function for patients > 70 years old
* Physical tests: walking speed and "hand grip" dynamometer secondary objectives:- Proposal of a composite score for the detection of sarcopenia usable in clinical routine
* Evaluation of nutritional intake
* Evaluation of the severity of undernutrition
* Verification of a correlation between the sarcopenia indices of ovarian and endometrial cancer
* Evaluate tolerance profiles to systemic treatments with regard to sarcopenia figures
* Assess the relationship between PFS, OS and sarcopenia index in cancer diagnosis secondary judgment criteria :
* Statistical analysis of sarcopenia and undernutrition data
* Quantification of ingestates (SEFI scale) +/- intake of oral nutritional supplement
* Serological tests: NFS, CRP and Albuminemia
* Comparison of sarcopenia index figures between ovarian and endometrial cancer
* Collection of the grades of toxicities and adverse events to systemic treatments in parallel with the measurement of sarcopenia.
* Correlation between progression-free survival, death and sarcopenia index at cancer diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patient presenting with a diagnosis of cancer of ovarian origin with an indication for chemotherapy
* Patient with a diagnosis of endometrial cancer with an indication for chemotherapy
* Patient with no diagnosis of other types of cancer in the previous five years
* Collection of consent
* Patient affiliated to a Social Security scheme

Exclusion Criteria:

* Patient with cancer of ovarian origin not requiring chemotherapy treatment
* Patient with endometrial cancer not requiring chemotherapy treatment
* Discovery of an intercurrent cancer other than skin or cervix cancers.
* Patient wearing a Pace maker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
clinical screening for sarcopenia | 36 month
  Identify the criteria correlated with the presence of sarcopenia (defined by the measurement of the IMS by the CT-X method in L3) among the impedancemetry and the HAS malnutrition criteria.
Proposal of a composite score for the detection of sarcopenia usable in clinical routine | 36 month
  Statistical analysis of sarcopenia and undernutrition data

CONTACTS AND LOCATIONS:
Overall Officials: fillon aurélie, Principal Investigator — Centre Hospitalier Metropole Savoie
Locations (1):
- Centre Hospitalier Metropole Savoie, Chambéry, Savoie, France

IPD SHARING:
Plan to Share IPD: No